CLINICAL TRIAL: NCT05710861
Title: Randomized Medical-Economic Trial Comparing Focal HIFU Treatment to Total Prostatectomy in Patients With Intermediate Prognosis Prostate Cancer
Brief Title: Cost-utility of Focal HIFU vs Prostatectomy
Acronym: EMERHIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHUBX 2019/67
Record Dates: First submitted 2023-01-16; First posted 2023-02-02 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
Keywords: Localized Prostate cancer; Prostatectomy; Focal HIFU; Quality of life; Cost; ISUP 2
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Multicentric pragmatic clinical trial, comparative, with no insu, randomized in two parallel groups with a 1:1 allocation ratio
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- F-HIFU Group (Experimental): 50 to 75 years old patients fit for a Radical Prostatectomy when active surveillance is not recommended and who do not want a radiation therapy: harboring a non-treated localized PC, with a maximum Gleason score of 3+4 , ISUP 2 and less than 50% of positive prostate biopsy (favorable intermediate risk), with or without contralateral microfocus score 3+3 (ISUP 1) of less than 3 mm, with a tumor visible on MRI and biopsy-proven with systematic and targeted biopsy with at least 2 biopsies per target and 12 systematic biopsies, Tumor involving maximum 2 biopsy-proven contiguous sextants. Patients with multiple MRI targets may be included if only one target is biopsy-proven, T1c-T2 stage, PSA <20 ng/ml, prostate volume less than 100 ml, fully informed patient accepting, after a decent reflexion time, to participate to the study by signing a consent form, affiliated or beneficiary patient to the French social security system
  Interventions: Device: F-HIFU
- Prostatectomy Group (Active Comparator): 50 to 75 years old patients fit for a Radical Prostatectomy when active surveillance is not recommended and who do not want a radiation therapy: harboring a non-treated localized PC, with a maximum Gleason score of 3+4 , ISUP 2 and less than 50% of positive prostate biopsy (favorable intermediate risk), with or without contralateral microfocus score 3+3 (ISUP 1) of less than 3 mm, with a tumor visible on MRI and biopsy-proven with systematic and targeted biopsy with at least 2 biopsies per target and 12 systematic biopsies, Tumor involving maximum 2 biopsy-proven contiguous sextants. Patients with multiple MRI targets may be included if only one target is biopsy-proven, T1c-T2 stage, PSA <20 ng/ml, prostate volume less than 100 ml, fully informed patient accepting, after a decent reflexion time, to participate to the study by signing a consent form, affiliated or beneficiary patient to the French social security system
  Interventions: Procedure: Radical Prostatectomy

INTERVENTIONS:
Device: F-HIFU — A F-HIFU treatment will be performed with the Focal-One® machine according to the predefined treatment area for each patient using the standard procedure in place in each therapeutic center and according to the user's manual edited by the company, under locoregional or general anaesthesia.
  Arms: F-HIFU Group
Procedure: Radical Prostatectomy — A Radical Prostatectomy will be performed according to the standard procedure in place in each center, under general anaesthesia, through an open, laparoscopic or robot-assisted laparoscopic approach
  Arms: Prostatectomy Group

SUMMARY:
Medico-Economic Randomized Trial comparing Focal HIFU Treatment to Radical Prostatectomy in Patients with Favorable Intermediate Risk Prostate Cancer

DETAILED DESCRIPTION:
Standard treatment option of intermediate risk (ISUP2) prostate cancer (PC) is either radical prostatectomy (RP) or radiation therapy (RT). An attractive option for selected patients and for the health care system would be to spare the preserved gland to decrease urinary, sexual and digestive side effects of whole-gland treatments keeping with a good cancer control. For these reasons, focal treatments have been developed in localized PC. The principal objective of the EMERHIT study is to estimate, from the health system point of view, the efficiency (cost/utility study) of focal HIFU (F-HIFU) for intermediate risk PC compared to RP (either by open, laparoscopic or robotic surgical approach) at 24 months. It will be a multicentric pragmatic clinical trial, comparative, with no insu, randomized in two parallel groups :

* (1) F-HIFU treatment
* (2) RP Randomization will be equal (ratio 1:1), stratified on the centers and performed maximum at 2 months before the procedure. The comparison to the SNDS data will use the NIR of the patients selected for the study. The use of the SNDS data will allow, on top of the estimation of the care cost, to increase the patient's follow-up (with no supplemental visit) and measure, at 48 months, costs, mortality rate and cancer control measures From version 4.0 of the protocol, randomisation will be adjusted to a 2:1 ratio and stratified by centre.

ELIGIBILITY:
Inclusion Criteria:

* 45-75 yo male harboring a non-treated localized prostatic adenocarcinoma of maximum Gleason score 3+4, ISUP 2 unilateral on at most maximum 2 contiguous sextants (favorable intermediate risk),with or without ipsilateral or contralateral focus of score 3+3 (ISUP1).
* Tumor visible on MRI and proven by systematic and/or targeted biopsies according to the center's practices, regardless of the route used (transrectal or transpirenal)
* Or patients under active surveillance whose follow-up prostate biopsies reveal unilateral ISUP2 on at most 2 contiguous sextants (favorable intermediate risk), with or without ipsilateral or contralateral Gleason 3+3 focus (ISUP1)
* Patients with several suspicious foci on MRI may be be included if only one of these foci is confirmed by targeted biopsies with an ISUP2 score. If more than one suspected site on MRI is confirmed by targeted biopsies, these should be unilateral ISUP2 on a maximum of 2 contiguous sextants (favourable intermediate risk), with or without an ipsilateral or contralateral site with a Gleason score of 3+3 (ISUP1).
* stage T1c-T2,
* with PSA <20 ng/ml,
* with prostate volume less than 150 ml,
* patient clearly informed of the study and having agreed, with sufficient time for reflection to participate by signing the study's informed consent form,
* patient affiliated to or benefiting from a social security scheme

Exclusion Criteria:

* Metastatic prostate cancer.
* Gleason score > 3+4 (ISUP>2).
* Adenoma prostate carcinoma Cribriform or intraductal.
* Previous treatment anterior for the same cancer, whatever modality.
* Contra-indication to pelvic MRI with gadolinium injection.
* Contra-indication to surgery or general anesthesia.
* Patient who refuse the one-year follow-up control biopsy after F-HIFU.
* Presence of implant (stent, catheter) less than 1 cm from the treatment area.
* Urinary or rectal fistula.
* Anal or rectal stenosis or any other abnormality that may interfere with the Focal One® endorectal probe introduction.
* Anatomic abnormality of the rectum or rectal mucosa.
* Presence of a urinary artificial sphincter, a penile prosthesis or intraprostatic implant, i.e. urethral prosthesis.
* Bladder neck and/or urethral stenosis or sclerosis.
* Inflammatory bowel disease (colon or rectum).
* Ongoing UTI (should be treated before the F-HIFU or the RP).
* Previous anal or rectal surgery that may interfere with the anal probe introduction.
* Latex allergy.
* Rectal wall thickness > 10 mm.
* Tumor not accessible to a F-HIFU treatment (tumors located in the fibro-muscular anterior zone).
* Previous not controlled cancer and/or treated since less than 5 years (except basocellular skin cancer).
* Patient not able to understand the trial objectives or refusing to adhere to the trial instructions.
* Patients under law-protection.
* Patient in an ongoing research trial.
* Patient with a severe health or psychologic problem that could impair the protocol pathway.

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2028-06-22 (Estimated); Study Completion 2028-06-22 (Estimated)

PRIMARY OUTCOMES:
The cost/utility ratio expressed as differential cost per QALY in favor of F-HIFU compared to RP (open, lap or robot) at 24 months. | 24 months
  Utility will be measured at baseline and at 6, 12 and 24 months using the EQ-5D-5L self-administered questionnaire.
  Costs will be estimated from the perspective of the French health system. They will be collected by probabilistic matching with data from the SNDS using data from the inclusion hospitalization of each patient included in the the trial.

SECONDARY OUTCOMES:
The per-year of preserved life differential cost between F-HIFU and RP | 48 months
  The per-year of preserved life differential cost at 48 months between F-HIFU and RP from the SNDS database evaluated by micro-costing
Differential cost between F-HIFU and open, lap or robotic RP | 24 months
  Differential cost of per-QALY improved at 24 months between F-HIFU and open, lap or robotic RP evaluated by micro-costing
Real production cost (€) of F-HIFU and RP | 48 months
  Real production cost (€) of F-HIFU and RP evaluated by micro-costing
Net benefit (€) for the Health Insurance | 48 months
  Net benefit (€) for the Health Insurance of a diffusion of F-HIFU into the French Health System for patients with favorable intermediate risk PC evaluated by micro-costing
Survival with no salvage treatmente. | 12, 24 and 48 months
  Survival with no salvage treatment at 12, 24 and 48 months, evaluated in part from the SNDS database. Optional salvage treatments possibly being: a second F-HIFU, RP or radiotherapy with or without androgen deprivation. All salvage treatments, except the F-HIFU, are already reimbursed by the French Health System and available in the SNDS database.
Overall survival | 12, 24 and 48 months
  Overall survival at 12, 24 and 48 months measured from the inclusion date to the date of death, all causes of death being included or the date of the last visit or at 48 months
Cancer specific survival | 12, 24 and 48 months
  Cancer specific survival at 12, 24 and 48 month measured from the date of inclusion to the date of death due to the progression of PC or the date of the last visit. Causes of death are available in the SNDS database since it is implemented by the CEpiDC
Androgen deprivation-free survival | 12, 24 and 48 months
  Androgen deprivation-free survival (equivalent to metastasis-free survival) at 12, 24 and 48 month measured from the inclusion date to the first prescription of androgen deprivation therapy or the date of the last visit
Urinary and sexual functions | Inclusion and 1, 6, 12 and 24 months
  Urinary and sexual functions will be evaluated at inclusion then at 6, 12 and, 24 month using auto-questionnaires EPIC-26
Patient's quality of life | Inclusion and 1, 6, 12 and 24 months
  Patient's quality of life will be evaluated at inclusion then at 6, 12 and 24 month using the auto-questionnaires EORTC QLQ C30
Urinary and sexual functions | Inclusion and 1, 6, 12 and 24 months
  Urinary and sexual functions will be evaluated at inclusion then at 6, 12 and, 24 month using auto-questionnars IPSS
Urinary and sexual functions | Inclusion and 1, 6, 12 and 24 months
  Urinary and sexual functions will be evaluated at inclusion then at 6, 12 and, 24 month using auto-questionnaires IIEF-5
Patient's quality of life | Inclusion and 1, 6, 12 and 24 months
  Patient's quality of life will be evaluated at inclusion then at 6, 12 and 24 month using the auto-questionnaires QLQ PR25
Patient's quality of life | Inclusion and 1, 6, 12 and 24 months
  Patient's quality of life will be evaluated at inclusion then at 6, 12 and 24 month using the auto-questionnaires EQ-5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Franck BLADOU, PROF, Principal Investigator — University Hospital, Bordeaux
Locations (20):
- France (19):
  - Clinique Saint Vincent, Besançon
  - Clinique Tivoli, Bordeaux
  - CHU de Bordeaux, Bordeaux
  - Hopitaux civil de Colmar, Colmar
  - CHU Grenoble Alpes, Grenoble
  - Hopital prive drome ardeche, Guilherand-Granges
  - Hopital Claude HURIEZ, Lille
  - Hopital Privé La Louviere, Lille
  - Hopital Edouard Herriot Pavillon V, Lyon
  - APHM Nord Marseille, Marseille
  - Hopital Cochin, Paris
  - Hopital Privé francheville, Périgueux
  - Hopital Lyon Sud HCL Bat 3C Centre, Pierre-Bénite
  - Clinique La Croix du Sud, Quint-Fonsegrives
  - CHU de Rennes, Rennes
  - CH Saintonge, Saint-Jean-d'Angély
  - Clinique Saint Michel, Toulon
  - CHU Toulouse rangueil, Toulouse
  - Clinique Oceane, Vannes
- CHU Pointe à Pitre, Pointe-à-Pitre, Guadeloupe